CLINICAL TRIAL: NCT03219151
Title: A Mixed-methods Evaluation of a Gamified Electronic Medication Administration Record (eMAR) System for Use in the Simulated Nursing Education
Brief Title: Evaluation of a Gamified Electronic Medication Administration Record (eMAR) System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: eCampusOntario (Unknown); Centre for Addiction and Mental Health (Other); Texas Tech University Health Sciences Center (Other); London Health Sciences Centre (Other); St. Joseph's Health Care London (Other); Wilfrid Laurier University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RI-WEST03
Record Dates: First submitted 2017-06-06; First posted 2017-07-17 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2017-05

CONDITIONS: Nurse's Role; Medication Administered in Error; Simulation of Physical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eMAR game (Experimental): Participants provided access to eMAR simulator game in advance of simulated return-demonstration; also receive normal education pre-work related to eMAR administration
  Interventions: Device: eMAR game; Other: Normal pre-work
- Normal pre-work (Active Comparator): Participants receive normal education pre-work related to eMAR administration, in advance of simulated return-demonstration
  Interventions: Other: Normal pre-work

INTERVENTIONS:
Device: eMAR game — The eMAR simulator videogame affords students a virtual and immersive opportunity to practice medication administration using an eMAR system, in a structured fashion that provides real-time feedback related to best-practices and safety compliance of the medication process
  Arms: eMAR game
Other: Normal pre-work — Participants complete normal education pre-work related to eMAR administration, in advance of simulated return-demonstration

SUMMARY:
This research project will evaluate a gamified electronic medication administration record (eMAR) system simulator as a mechanism to improve students' learning of medication administration in simulated clinical education. The gamified eMAR simulator will be evaluated using a pragmatic randomized controlled trial design in order to determine the effectiveness of the game as a technology-enabled, online learning intervention.

DETAILED DESCRIPTION:
The main objective of this study is to examine whether the use of a gamified medication administration simulator improves nursing students' medication administration safety within simulated practice; increases student self-efficacy and knowledge of the medication administration process; and, improves motivational and cognitive processing attributes related to student learning in a technology-enabled environment. It is hoped that by completing this trial, the effectiveness of using an eMAR simulator as an educational tool to better prepare nursing students to administer medications using eMAR technology for practice will be ascertained.

ELIGIBILITY:
Inclusion Criteria:

* (1) second year nursing students; and, (2) partaking in clinical simulated education in either in Fall 2017 or Winter 2018 semesters.

Exclusion Criteria:

* (1) A student who is not enrolled the BScN program at the respective site of data collection, in Fall 2017 or Winter 2018.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Frequency of medication errors | weeks 6-9
  Number medication errors generated by nursing students, as assessed by a previously modified researcher-developed rubric that assists observers to quantify the number of medication errors generated during a return-demonstration in clinical simulation (DOI:10.1097/NNE.0000000000000361 / 10.1016/j.ecns.2017.05.016). The quantity of medication errors are codified in six categories: infection control; assessment; verification; scan; administration; documentation.

SECONDARY OUTCOMES:
Self-efficacy of eMAR medication administration instrument | weeks 4-9
  Self-efficacy of eMAR medication process will be assessed through a pre/post survey. The scale is 6 item scale (1=not confident; 7=absolutely confident). The higher the index, the higher an individual's perceived self-efficacy toward eMAR medication administration. Used as a pre/post test, this instrument will measure changes over time related to eMAR medication administration self-efficacy
Game motivational and cognitive attributes of participants instrument | week 9
  Cross-sectional data will be collected using questions modified from the Huang et al. (2011) validated instrument that measures motivational (i.e., attention, relevance, confidence, satisfaction) and cognitive processing of learning in technology-enabled environments (20 questions, Cronbach's alpha = 0.91). This composite outcome is reported through tests of dimensionality, using a canonical correlational analysis, providing standardized coefficients between the instrument's sub-components.
Knowledge of eMAR medication administration instrument | weeks 4-9
  Knowledge of eMAR medication process will be assessed through a pre/post survey. The scale is 8 item scale (1=not prepared; 7=absolutely prepared). The higher the index, the higher an individual's perceived knowledge toward eMAR medication administration. Used as a pre/post test, this instrument will measure changes over time related to eMAR medication administration knowledge

CONTACTS AND LOCATIONS:
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Booth R, Sinclair B, McMurray J, Strudwick G, Watson G, Ladak H, Zwarenstein M, McBride S, Chan R, Brennan L. Evaluating a Serious Gaming Electronic Medication Administration Record System Among Nursing Students: Protocol for a Pragmatic Randomized Controlled Trial. JMIR Res Protoc. 2018 May 28;7(5):e138. doi: 10.2196/resprot.9601. PMID 29807885